CLINICAL TRIAL: NCT04795310
Title: A Clinical Observation on the Efficacy and Safety of Pulsed Dye Laser and Intense Pulsed Light With Different Wavelength Bands in the Treatment of Facial Telangiectasia: a Retrospective, Self-controlled Trial
Brief Title: Clinical Observation of Pulsed Dye Laser and Intense Pulsed Light in Treating Facial Telangiectasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, Gang Wang, Chief of Dermatology, Xijing Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XijingH-PF-20192074-C-1
Record Dates: First submitted 2019-07-02; First posted 2021-03-12 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: Telangiectasia
Keywords: Facial Telangiectasia; Pulsed dye laser (PDL); Intense Pulsed Light
MeSH Terms: conditions — Telangiectasis | interventions — Lasers, Dye; Intense Pulsed Light Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pulsed Dye Laser (Experimental): PDL (Vbeam perfecta, 595 nm, Candela Corporation, Wayland, MA) was used with energy dosages of 9-11J/cm2, pulse durations of 10ms/20ms, and 7 or 10 mm handpieces with dynamic cooling device (DCD)
  Interventions: Device: Pulsed dye laser
- Intense Pulsed Light (Active Comparator): Vascular wavelength bands of 530-650nm and 900-1200nm
  Interventions: Device: Pulsed dye laser

INTERVENTIONS:
Device: Pulsed dye laser — PDL (Vbeam perfecta, 595 nm, Candela Corporation, Wayland, MA) was used with energy dosages of 9-11J/cm2, pulse durations of 10ms/20ms, and 7 or 10 mm handpieces with dynamic cooling device (DCD).
  IPL device (M22, Lumenis Limited, Yokneam, Israel) with integration of sapphire ChillTip system for epidermal cooling were used in the study. Three wavelength bands were configured: 560-1200 nm, 590-1200 nm, and vascular wavelength bands of 530-650nm and 900-1200nm. All the treatment handpieces had a spot size of 15mm×35mm, fluence of 9-17J/cm², pulse duration of 4.0-6.0ms and pulse delay of 20-40ms, underwent the M22 advanced optimal pulse technology (AOPT) treatment.
  Other Names: Intense pulsed light

SUMMARY:
1. Facial telangiectasia is one of the common skin vascular lesions characterized by dilated cutaneous vasculatures in the skin surface or mucous membranes. Lesions are generally sensitive to exposure of cold, heat and sun. Those distinct small dilated blood vessels are cosmetically disfiguring for patients which require an effective solution. The traditional management options for facial telangiectasia include cryotherapy, CO2 laser, topical agent, oral estrogens, electrosurgery, and radioactive treatment. However, inadequate outcomes and severe adversaries are the major concerns to patients and physicians.
2. Pulsed dye laser (PDL) is effective for vasodilatory diseases, especially for the superficial to middle layers of the dermis.

   The intense pulsed light source is an alternative or supplement to the already existing laser devices that are part of the laser surgeon's repertoire. The broad wavelength spectrum and variable pulse duration allow greater penetration depths to be reached without damaging surrounding tissue and thus enhance the versatility of this system.
3. This study aims to compare the clearance efficacy of facial telangiectasia using PDL (595nm) with IPL configured by various wavelength bands, including M22 vascular filter (530-650nm and 900-1200nm), M22 560 (560-1200nm), M22 590 (590-1200nm) .

DETAILED DESCRIPTION:
Detailed Description has not been entered.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be clinically diagnosed with facial telangiectasia
* No other external treatment was performed before the injury was treated

Exclusion Criteria:

* subjects with a recent history of exposure to sunlight
* subjects allergic to topical anesthesia
* subjects with scar constitution
* subjects with skin malignant tumors or precancerous lesions
* subjects with diabetes, heart disease, epilepsy, connective tissue disease, etc
* subjects who Pregnant or breast feeding
* subjects with recent skin infections (such as viruses, bacteria, etc.)
* other methods are being used to treat subjects with similar diseases
* subject who have taken isotretinoin A in the past year
* subject with facial dermatitis

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Severity index of facial telangiectasia | 6months
  1. minimal, focal visible telangiectasia in 5-10% of anatomic area
  2. focal visible telangiectasia in11-20% of an anatomic area
  3. focal visible telangiectasia in 21-30% of anatomic area
  4. visible telangiectasia in 31-40% of anatomic area
  5. visible telangiectasia in 41-50% of anatomic area
  6. moderately severe telangiectasia in 51-60% of anatomic area
  7. moderately severe telangiectasia in 61-70% of anatomic area
  8. severe telangiectasia in 71-80% of anatomic area
  9. severe telangiectasia in 81-90% of anatomic area
  10. severe and diffuse facial telangiectasia in entire anatomic area for facial telangiectasia

CONTACTS AND LOCATIONS:
Overall Officials: Gang Wang, Prof, Principal Investigator — Dermatology Derpartment of Xijing Hospital
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China